CLINICAL TRIAL: NCT02307279
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Assessing the Effect of Gelesis100 on Body Weight in Overweight and Obese Subjects With and Without Type 2 Diabetes
Brief Title: Study of Gelesis100 on Body Weight in Overweight and Obese Subjects With and Without Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gelesis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G-04
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Gelesis100 (Experimental): Gelesis100 twice daily
  Interventions: Device: Gelesis100
- Placebo (Placebo Comparator): Matching placebo twice daily
  Interventions: Device: placebo

INTERVENTIONS:
Device: Gelesis100
  Arms: Gelesis100
Device: placebo
  Arms: Placebo

SUMMARY:
This study will asses the decrease in body weight after repeated administration of Gelesis100 in overweight and obese subjects with and without Type 2 Diabetes.

DETAILED DESCRIPTION:
To asses the decrease in body weight after repeated administration of Gelesis100 in overweight and obese subjects with and without Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 to 65 years of age, inclusive
* Signed Informed Consent Form
* BMI 27 to 40, inclusive (BMI of <30 should have at least one comorbidity)
* Fasting plasma glucose 90mg/dL to 145 mg/dL, inclusive; non-diabetic normoglycemic (fasting glucose 90 mg/dL to 100 mg/dL, inclusive); non-diabetic impaired fasting glucose 100mg/dL to 126 mg/dL; and diabetic: untreated (126 mg/dL to 145 mg/dL, inclusive) and metformin-treated (metformin dose 1500mg/DL and less, fasting glucose less than 145 mg/dL, inclusive)

Exclusion Criteria:

* Pregnancy or lactation
* Absence of medically approved contraceptive methods in females of childbearing potential
* History of allergic reaction to modified cellulose, citric acid, sodium stearyl fumarate, raw cane sugar, gelatin, and titanium oxide
* Administration of investigational products within 1 month prior to Screening Visit
* Subjects who stopped smoking within 6 months prior to Screening Visit or considering smoking cessation during the study
* Subjects anticipating surgical intervention during the study
* Known Type 1 diabetes
* History of eating disorders
* Angina, coronary bypass, or myocardial infarction within 6 months prior to Screening Visit
* History of: swallowing disorders, esophogeal anatomic abnormalities, gastroesophageal reflux disease, gastric or duodenal ulcer, gastroparesis (chronic nausea, vomiting, heartburn...), gastric bypass or other gastric surgery, intestinal obstruction or at high risk of including suspected small bowel adhesion, pancreatitis, malabsorption, history of bowel resection (except if related to appendectomy), history of abdominal radiation treatment
* Laxative users
* History of: HIV, hepatitis B or C; cancer within the past 5 years
* Abnormal serum thyroid-stimulating hormone (TSH)
* Positive urine drug test
* Anti-obesity medication within 1 month prior to Screening Visit (except stable doses of metformin, no more than 1500 mg/day, for at leaset 1 month in subjects with type 2 diabetes)
* Systemic corticosteroids within 1 month prior to Screening Visit
* Thyroid hormones or preparations within 1 month prior to Screening Visit
* Estrogen within 1 month prior to Screening Visit
* Any other medication known to cause weight loss or weight gain within 1 month prior to Screening Visit
* TSH suppression therapy for thyroid cancer
* medications requiring mandatory administration with meal (lunch or dinner), except metformin
* Other medication or product used for chronic diseases if their impaired gastrointestinal absorption can cause safety issues
* Change in medications treating hypertension and/or dyslipidemia within 1 month prior to Screening Visit (including change in dose)
* Anticipated requirement for use of prohibited concomitant medication

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan M Heshmati, MD, Study Director — Chief Medical Officer
Locations (33):
- United States (24):
  - Investigative Site, Anaheim, California
  - Investigative Site, San Diego, California
  - Investigative Site, Tustin, California
  - Investigative Site, Walnut Creek, California
  - Investigative Site, West Hills, California
  - Investigative Site, Aurora, Colorado
  - Investigative Site, Jacksonville, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, Boise, Idaho
  - Investigative Site, Chicago, Illinois
  - Investigative Site, Baton Rouge, Louisiana
  - Investigative Site, Boston, Massachusetts
  - Investigative Site, Las Vegas, Nevada
  - Investigative Site, New York, New York
  - Investigative Site, Raleigh, North Carolina
  - Investigative Site, Cincinnati, Ohio
  - Investigative Site, Columbus, Ohio
  - Investigative Site, Danville, Pennsylvania
  - Investigative Site, Nashville, Tennessee
  - Investigative Site, Dallas, Texas
  - Investigative Site, Round Rock, Texas
  - Investigative Site, West Jordan, Utah
  - Investigative Site, Norfolk, Virginia
  - Investigative Site, Richmond, Virginia
- Canada (2):
  - Investigative Site, Ottawa, Ontario
  - Investigative Site, Québec, Quebec
- Czechia (2):
  - Investigative Site, Hradec
  - Investigative Site, Prague
- Investigative Site, Copenhagen, Denmark
- Italy (3):
  - Investigative Site, Milan, Milanese
  - Investigative Site, Naples
  - Investigative Site, Rome
- Investigative Site, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Gelesis100: Gelesis100 twice daily
  Gelesis100
- Placebo: Matching placebo twice daily
  placebo
Period: Overall Study
Arm/Group | Gelesis100 | Placebo
Started | 223 | 213
Completed | 172 | 152
Not Completed | 51 | 61

BASELINE CHARACTERISTICS:
Population: All 436 randomized subjects were included in the ITT population and 434 (99.5%) subjects were included in the Safety Population. Two randomized subjects never received IP and were excluded from the Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gelesis100 | Placebo | Total
Number analyzed (Participants) | 223 | 213 | 436
Age, Categorical [Count of Participants; unit: Participants] — The age inclusion criteria used was ≥ 22 years and ≤ 65 years.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 223 | 213 | 436
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — All male and female ambulatory subjects who met all inclusion criteria and no exclusion criteria were allowed to participate in the study.
  Participants
    Female | 125 | 120 | 245
    Male | 98 | 93 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ambulatory subjects who met all inclusion criteria and no exclusion criteria were allowed to participate in the study regardless of ethnicity
  Participants
    Hispanic or Latino | 11 | 16 | 27
    Not Hispanic or Latino | 212 | 197 | 409
    Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ambulatory subjects who met all inclusion criteria and no exclusion criteria were allowed to participate in the study regardless of race/ethnicity.
  Participants
    White | 189 | 180 | 369
    Black or African American | 26 | 24 | 50
    Asian | 4 | 4 | 8
    Other | 2 | 5 | 7
    American Indian or Alaska Native | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Europe | 126 | 119 | 245
  United States | 97 | 94 | 191

OUTCOME MEASURES:

1. Primary Outcome: Co-Primary Outcome: Percent Change in Body Weight
Description: Percent change in body weight from Baseline to Day 171 is presented.
Time Frame: Baseline to Day 171
Population: Overall number of patients analyzed is equal to the intention to treat population (all randomized subjects).
Measure: Mean (Standard Deviation); unit: percentage change in body weight
Arm/Group | Gelesis100 | Placebo
Number analyzed (Participants) | 223 | 213
percentage change in body weight | -6.41 (5.79) | -4.39 (5.52)
Statistical Analysis 1: Comparison: Gelesis100 vs Placebo; Simple Superiority, H0: μ (Placebo) -μ (Gelesis100) = 0; Test type: Superiority; p = 0.0007, ANCOVA; Adjusted for stratification factors, and baseline weight; Mean Difference (Net) = -2.07, 95% CI 2-sided [-3.24 to -0.90], Standard Error of Mean 0.59 — Difference in adjusted mean taken for comparability between the two groups (treatment - placebo)
Statistical Analysis 2: Comparison: Gelesis100 vs Placebo; Super-Superiority (>3% difference), H0: μ(Placebo)-μ(Gelesis100) < 3%; Test type: Superiority; p = 0.1193, ANCOVA; Adjusted for stratification factors, and baseline weight

2. Primary Outcome: Co-Primary Outcome: Percentage of Subjects Who Achieve Body Weight Loss ≥ 5%
Description: Percentage of participants who achieve a body weight loss ≥ 5% from Baseline to Day 171 is presented.
Time Frame: Baseline to Day 171
Population: Overall Number of Participants Analyzed is equal to the intention to treat population (all randomized subjects).
Measure: Number; unit: percentage of participants
Arm/Group | Gelesis100 | Placebo
Number analyzed (Participants) | 223 | 213
percentage of participants | 58.6 | 42.2
Statistical Analysis 1: Comparison: Gelesis100; H0: π (Gelesis100)< 0.35; Test type: Superiority — The performance goal for body weight responders was set at 35%; p < 0.0001, Binomial Proportion Test
Statistical Analysis 2: Comparison: Gelesis100 vs Placebo; OR-trt refers to the odds ratio of being a body weight responder for Gelesis100 vs. Placebo. H0: OR-trt= 1; Test type: Superiority; p = 0.0008, Regression, Logistic; Adjusted for stratification factors and baseline weight; Odds Ratio (OR) = 2.01, 95% CI 2-sided [1.34 to 3.01]

3. Secondary Outcome: Percent Body Weight Change in Subjects With Impaired Plasma Glucose Status at Baseline
Description: Impaired plasma glucose status is defined as Fasting Plasma Glucose (FPG) ≥100mg/dL and <126mg/dL at baseline measurement.
Time Frame: Baseline to Day 171
Population: Overall Number of Participants Analyzed is equal to the number of participants with impaired fasting glucose at Baseline.
Measure: Mean (Standard Deviation); unit: percentage change in body weight
Arm/Group | Gelesis100 | Placebo
Number analyzed (Participants) | 59 | 58
percentage change in body weight | -6.46 (6.28) | -5.54 (6.08)

4. Secondary Outcome: Change in Plasma Glucose Status (Normal, Impaired, Diabetic) in Subjects With Impaired Plasma Glucose Status at Baseline.
Description: Normal plasma glucose status is defined FPG ≤ 100mg/dL. Impaired plasma glucose status is defined as FPG ≥100mg/dL and <126mg/dL. Diabetic plasma glucose status was defined as FPG >126mg/dL.
Time Frame: Baseline to Day 171
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Gelesis100 | Placebo
Number analyzed (Participants) | 59 | 58
participants
  Normal | 23 | 19
  Impaired (Pre-diabetic) | 35 | 34
  Diabetic | 1 | 5

5. Secondary Outcome: Percent Change in Plasma Glucose
Description: Percent change in Plasma Glucose in subjects with impaired glucose and T2D at baseline. Impaired plasma glucose is defined as FPG≥100mg/dL and FPG<126mg/dL.
Time Frame: Baseline to Day 171
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of change in plasma glucose
Arm/Group | Gelesis100 | Placebo
Number analyzed (Participants) | 59 | 58
percentage of change in plasma glucose | -2.39 (20.55) | -1.95 (14.61)

6. Secondary Outcome: Change in Body Mass Index (BMI)
Description: The BMI was calculated using height (in cm) and weight (in kg) according to the following formula: BMI (kg/m2((superscript 1)) = Weight (kg)/[Height (cm)/100]2(superscript2).
Time Frame: Baseline to Day 171
Population: Overall number of patients analyzed is equal to the number of all participants with available data.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Gelesis100 | Placebo
Number analyzed (Participants) | 223 | 213
kg/m^2 | -2.12 (1.92) | -1.51 (1.90)

7. Secondary Outcome: Change in Hemoglobin HbA1c in Subjects With Type 2 Diabetes at Baseline
Description: To assess the decrease in HbA1c after repeated administration of Gelesis 100 over a period of 168 days in overweight and obese people with type 2 diabetes, The glycosylated hemoglobin was measured in mmol/mol.
Time Frame: Baseline to Day 171
Population: Overall number of patients analyzed is equal to the number of all participants with type 2 diabetes at baseline.
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Gelesis100 | Placebo
Number analyzed (Participants) | 21 | 25
mmol/mol | -0.64 (5.07) | -3.06 (4.18)

8. Other Pre Specified Outcome: Assess Safety and Tolerability of Administration of Gelesis100
Description: Adverse Events (AEs), Physical Examinations, Vital Signs, Laboratory Tests
Time Frame: Baseline to Day 197
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From screening (Day -21) to Day 197. The adverse device effect (AE) and the serious adverse device effects (SAE) are collected since screening until 28 days after the last administration of the investigational medical device.
Description: AE reported by subjects are recorded and discussed in detail by the investigator at each visit.
Arm/Group | Gelesis100 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/223 | 0/211
Serious Adverse Events (participants affected / at risk) | 0/223 | 1/211
Other Adverse Events (participants affected / at risk) | 159/223 | 149/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gelesis100 (N=223) | Placebo (N=211)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gelesis100 (N=223) | Placebo (N=211)
Abdominal Distention (Gastrointestinal disorders) | 26 (27) | 14 (14)
Abdominal pain (Gastrointestinal disorders) | 12 (12) | 6 (6)
Constipation (Gastrointestinal disorders) | 12 (13) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 28 (31) | 18 (20)
Flatulence (Gastrointestinal disorders) | 19 (21) | 11 (14)
Infrequent bowel movements (Gastrointestinal disorders) | 21 (24) | 10 (12)
Nausea (Gastrointestinal disorders) | 11 (12) | 11 (12)
Nasopharyngitis (Infections and infestations) | 26 (31) | 30 (37)
Upper respiratory tract infections (Infections and infestations) | 8 (9) | 12 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 13 (13)
Headache (Nervous system disorders) | 16 (23) | 18 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT02307279/Prot_SAP_000.pdf